CLINICAL TRIAL: NCT03879174
Title: A Phase II Study of Pembrolizumab And Tamoxifen Among Women With Advanced Hormone Receptor Positive Breast Cancer And Esr1 Mutation
Brief Title: Pembrolizumab And Tamoxifen Among Women With Advanced Hormone Receptor Positive Breast Cancer And Esr1 Mutation
Acronym: Pembro
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mediclinic Middle East (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AN.MCME.CR.12; MISP # 55574 (Other: MSD Inc.)
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Breast Cancer Female
Keywords: HR Positive Breast Cancer
MeSH Terms: interventions — pembrolizumab; Tamoxifen

STUDY DESIGN:
Intervention Model Description: Recently there has been a growing interest in using immune check point inhibitors in breast cancer especially among patients with triple negative and HER2 positive subtypes that are thought to be more immunogenic compared to the luminal subtypes. However there has been a growing interest in looking at immune check point inhibitors among patients with hormone receptor positive breast cancer as a potential method of overcoming endocrine resistance. In the current study we propose a phase II trial to evaluate the anti-tumor activity of pembrolizumab and tamoxifen among patients with hormone receptor positive, HER2 negative metastatic breast cancer who have progressed on a prior aromatase inhibitor and have acquired an ESR1 mutation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab + Tamoxifen (Experimental): Pembrolizumab (200mg IV every three weeks) + Tamoxifen (20 mg OD)
  Interventions: Drug: Pembrolizumab + Tamoxifen

INTERVENTIONS:
Drug: Pembrolizumab + Tamoxifen — The choice of the 200 mg Q3W as an appropriate dose for the switch to fixed dosing is based on simulations performed using the population PK model of pembrolizumab showing that the fixed dose of 200 mg every 3 weeks will provide exposures that 1) are optimally consistent with those obtained with the 2 mg/kg dose every 3 weeks, 2) will maintain individual patient exposures in the exposure range established in melanoma as associated with maximal efficacy response and 3) will maintain individual patients exposure in the exposure range established in melanoma that are well tolerated and safe.
  A fixed dose regimen will simplify the dosing regimen to be more convenient for physicians and to reduce potential for dosing errors. A fixed dosing scheme will also reduce complexity in the logistical chain at treatment facilities and reduce wastage.

SUMMARY:
Pembrolizumab is a potent and highly selective humanized monoclonal antibody (mAb) designed to directly block the interaction between PD-1 and its ligands and enable the T cell to remain active and co-ordinate an attack on tumor cells.

We hypothesise that the Clinical Benefit Rate (CBR) and progression free survival (PFS) of metastatic breast cancer patients who have ESR1 mutation will improve following administration of a combination of pembrolizumab and tamoxifen.

DETAILED DESCRIPTION:
3.4.1 Pharmaceutical and Therapeutic Background The importance of intact immune surveillance in controlling outgrowth of neoplastic transformation has been known for decades. Accumulating evidence shows a correlation between tumor-infiltrating lymphocytes (TILs) in cancer tissue and favorable prognosis in various malignancies. In particular, the presence of CD8+ T-cells and the ratio of CD8+ effector T-cells / FoxP3+ regulatory T-cells seems to correlate with improved prognosis and long-term survival in many solid tumors.

The PD-1 receptor-ligand interaction is a major pathway hijacked by tumors to suppress immune control. The normal function of PD-1, expressed on the cell surface of activated T-cells under healthy conditions, is to down-modulate unwanted or excessive immune responses, including autoimmune reactions. PD-1 (encoded by the gene Pdcd1) is an Ig superfamily member related to CD28 and CTLA-4 which has been shown to negatively regulate antigen receptor signaling upon engagement of its ligands (PD-L1 and/or PD L2). The structure of murine PD-1 has been resolved. PD-1 and family members are type I transmembrane glycoproteins containing an Ig Variable-type (V-type) domain responsible for ligand binding and a cytoplasmic tail which is responsible for the binding of signaling molecules. The cytoplasmic tail of PD-1 contains 2 tyrosine-based signaling motifs, an immunoreceptor tyrosine-based inhibition motif (ITIM) and an immunoreceptor tyrosine-based switch motif (ITSM). Following T-cell stimulation, PD 1 recruits the tyrosine phosphatases SHP-1 and SHP-2 to the ITSM motif within its cytoplasmic tail, leading to the dephosphorylation of effector molecules such as CD3ζ, PKCθ and ZAP70 which are involved in the CD3 T-cell signaling cascade. The mechanism by which PD-1 down modulates T-cell responses is similar to, but distinct from that of CTLA-4 as both molecules regulate an overlapping set of signaling proteins. PD-1 was shown to be expressed on activated lymphocytes including peripheral CD4+ and CD8+ T-cells, B-cells, T regs and Natural Killer cells. Expression has also been shown during thymic development on CD4-CD8- (double negative) T-cells as well as subsets of macrophages and dendritic cells. The ligands for PD-1 (PD-L1 and PD-L2) are constitutively expressed or can be induced in a variety of cell types, including non-hematopoietic tissues as well as in various tumors. Both ligands are type I transmembrane receptors containing both IgV- and IgC-like domains in the extracellular region and contain short cytoplasmic regions with no known signaling motifs. Binding of either PD-1 ligand to PD-1 inhibits T-cell activation triggered through the T-cell receptor. PD-L1 is expressed at low levels on various non-hematopoietic tissues, most notably on vascular endothelium, whereas PD-L2 protein is only detectably expressed on antigen-presenting cells found in lymphoid tissue or chronic inflammatory environments. PD-L2 is thought to control immune T-cell activation in lymphoid organs, whereas PD-L1 serves to dampen unwarranted T-cell function in peripheral tissues. Although healthy organs express little (if any) PD-L1, a variety of cancers were demonstrated to express abundant levels of this T-cell inhibitor. PD-1 has been suggested to regulate tumor-specific T-cell expansion in subjects with melanoma (MEL). This suggests that the PD-1/PD-L1 pathway plays a critical role in tumor immune evasion and should be considered as an attractive target for therapeutic intervention.

Pembrolizumab is a potent and highly selective humanized monoclonal antibody (mAb) of the IgG4/kappa isotype designed to directly block the interaction between PD-1 and its ligands, PD-L1 and PD-L2. KeytrudaTM (pembrolizumab) has been approved in the United States for the treatment of patients with unresectable or metastatic melanoma and disease progression following ipilimumab and, if BRAF V600 mutation positive, a BRAF inhibitor. KeytrudaTM (pembrolizumab) is also a U.A.E. Ministry of Health registered medication.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible for participation in this trial, the subject must:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be 18 years of age on day of signing informed consent.
3. Have measurable disease based on RECIST 1.1.
4. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Sponsor.
5. Have a performance status of 0 or 1 on the ECOG Performance Scale.
6. Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 10 days of treatment initiation.

   Table 1 Adequate Organ Function Laboratory Values System Laboratory Value Hematological Absolute neutrophil count (ANC) ≥1,500 /mcL Platelets ≥100,000 / mcL Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment) Renal Serum creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 X upper limit of normal (ULN) OR

   ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN Hepatic Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR

   ≤ 5 X ULN for subjects with liver metastases Albumin >2.5 mg/dL Coagulation International Normalized Ratio (INR) or Prothrombin Time (PT)

   Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

   ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants aCreatinine clearance should be calculated per institutional standard.

9. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

10. Female subjects of childbearing potential (Section 5.7.2) must be willing to use an adequate method of contraception as outlined in Section 5.7.2 - Contraception, for the course of the study through 120 days after the last dose of study medication.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

The subject must be excluded from participating in the trial if the subject:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has a known history of active TB (Bacillus Tuberculosis)
4. Hypersensitivity to pembrolizumab or any of its excipients.
5. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
6. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
8. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
10. Has known history of, or any evidence of active, non-infectious pneumonitis.
11. Has an active infection requiring systemic therapy.
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
14. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
15. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
16. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
17. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
18. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | defined as time from enrollment to disease progression or death, whichever occurred first, assessed for a period of up to 36 months.
  time from enrollment to disease progression or death, whichever occurred first
Overall Response Rate (ORR) | Time for patient to achieve a complete response, partial response and stable disease in response to pembrolizumab therapy, assessed for a period of up to 36 months.
  percentage of patients with a best overall response of complete response (CR) or partial response (PR)

SECONDARY OUTCOMES:
Overall Survival | The length of time from the start of pembrolizumab treatment following which the patients are still alive, assessed for a period of up to 36 months.
  Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Dronsfield, Study Director — Hospital Director- Mediclinic City Hospital; Shaheenah Dawood, Principal Investigator — Consultant Oncologist
Locations (1):
- Mediclinic City Hospital, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baselga J, Campone M, Piccart M, Burris HA 3rd, Rugo HS, Sahmoud T, Noguchi S, Gnant M, Pritchard KI, Lebrun F, Beck JT, Ito Y, Yardley D, Deleu I, Perez A, Bachelot T, Vittori L, Xu Z, Mukhopadhyay P, Lebwohl D, Hortobagyi GN. Everolimus in postmenopausal hormone-receptor-positive advanced breast cancer. N Engl J Med. 2012 Feb 9;366(6):520-9. doi: 10.1056/NEJMoa1109653. Epub 2011 Dec 7. PMID 22149876
- [Background] Finn RS, Martin M, Rugo HS, Jones S, Im SA, Gelmon K, Harbeck N, Lipatov ON, Walshe JM, Moulder S, Gauthier E, Lu DR, Randolph S, Dieras V, Slamon DJ. Palbociclib and Letrozole in Advanced Breast Cancer. N Engl J Med. 2016 Nov 17;375(20):1925-1936. doi: 10.1056/NEJMoa1607303. PMID 27959613
- [Background] Toy W, Shen Y, Won H, Green B, Sakr RA, Will M, Li Z, Gala K, Fanning S, King TA, Hudis C, Chen D, Taran T, Hortobagyi G, Greene G, Berger M, Baselga J, Chandarlapaty S. ESR1 ligand-binding domain mutations in hormone-resistant breast cancer. Nat Genet. 2013 Dec;45(12):1439-45. doi: 10.1038/ng.2822. Epub 2013 Nov 3. PMID 24185512
- [Background] Rugo HS, Delord J-P, Im S-A, Ott PA, Piha-Paul SA, Bedard PL, Sachdev J, Le Tourneau C, van Brummelen E, Varga A, Saraf S, Pietrangelo D, Karantza V, Tan A.[S5-07] Preliminary efficacy and safety of pembrolizumab (MK-3475) in patients with PD-L1-positive, estrogen receptor-positive (ER+)/HER2-negative advanced breast cancer enrolled in KEYNOTE-028; Oral Session: General Session 5 (9:30 AM-11:30 AM); SABCS 2015
- [Background] Vonderheide RH, LoRusso PM, Khalil M, Gartner EM, Khaira D, Soulieres D, Dorazio P, Trosko JA, Ruter J, Mariani GL, Usari T, Domchek SM. Tremelimumab in combination with exemestane in patients with advanced breast cancer and treatment-associated modulation of inducible costimulator expression on patient T cells. Clin Cancer Res. 2010 Jul 1;16(13):3485-94. doi: 10.1158/1078-0432.CCR-10-0505. Epub 2010 May 17. PMID 20479064